CLINICAL TRIAL: NCT05901987
Title: A Multi-center, Open Label, Single-arm, Dose Ascending Clinical Trial for Evaluation of Safety and Efficacy of Gene Therapy Drug GC101 in the Treatment of Spinal Muscular Atrophy (SMA) Type 2 Patients
Brief Title: Evaluation of Safety and Efficacy of Gene Therapy Drug in the Treatment of Spinal Muscular Atrophy (SMA) Type 2 Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeneCradle Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JLJY-GC101-SMA-003
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: SMA II
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dosing group (Experimental): 1.2x10^14 vg/person of GC101 delivered one-time intrathecally (n=3)
  Interventions: Genetic: GC101
- Medium dosing group (Experimental): 2.4x10^14 vg/person of GC101 delivered one-time intrathecally (n=3)
  Interventions: Genetic: GC101
- High dosing group (Experimental): 4.8x10^14 vg/person of GC101 delivered one-time intrathecally (n=3)
  Interventions: Genetic: GC101

INTERVENTIONS:
Genetic: GC101 — Self-complementary AAV9 carrying a codon-optimized SMN coding sequence(coSMN1) driven by CMV enhancer and chicken β-actin promoter

SUMMARY:
The study will evaluate safety and efficacy of intrathecal delivery of GC101 gene therapy drug as a treatment of spinal muscular atrophy Type 2 (SMA 2) patients.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate safety and efficacy of gene therapy drug GC101 in SMA 2 patients. Open-label, dose-escalation clinical trial of GC101 will be conducted in multiple centers in China.

GC101 will be administrated intrathecally. Short-term safety will be evaluated in 52 weeks and enter long-term follow-up study of 5 years at will. Patients will be tested at baseline and followed up on various time points.

The primary analysis for efficacy will be assessed at 12 months after treatment with GC101 on the motor milestone of stand unassisted for at least 3 seconds for patients of age between 6 and 24 months, or changes from baseline HFMSE scores for patients of age between 24 and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 months and 60 months of age on day of signing informed consent form;
* Patient with SMA Type 2 as defined by the following features:

  * Diagnosis of SMA based on gene mutation analysis with bi-allelic SMN1 mutations (deletion or point mutations) and 2 copies of SMN
  * Onset of disease between 6 and 18 months of age
* Patient who can sit alone but never be able to stand or walk alone ;
* The patient's legal guardian(s) must be able to understand the purpose and risks of the study and voluntarily provide signed and dated informed consent prior to any study-related procedures being performed.

Exclusion Criteria:

* Patient who has participated in any previous gene therapy research trials;
* Patient who has received Nusinersen within 4 months and Risdiplam within 15 days before treatment;
* Patient who has AAV9 neutralizing antibody titer ≥1:200;
* Patient with a point mutation in SMN2 (c.859G>C);
* Patient who requires non-invasive ventilatory support averaging≥12 hours/day at screening, or use invasive ventilatory support or pulse oximetry < 95% saturation while awake and calm at screening;
* Patient who is positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis C antibody, or treponema pallidum antibody;
* Abnormal laboratory values considered clinically significant, including gamma-glutamyl transferase(GGT), Aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin > 3x upper limit of normal (ULN), Hemoglobin (Hgb)< 110 or >150 g/L, platelet <lower limit of normal (LLN);Class IV patient based on Modified Ross Heart Failure Classification for Children;
* Patient with a history of glucocorticoid allergy;
* Contraindication that would interfere with the lumbar puncture procedures;
* Presence of an untreated active infection requiring systemic antiviral therapy at any time during the screening period;
* Vaccination less than 2 weeks before infusion of vector;
* Patient who has any concurrent clinically significant major disease or any other condition that, in the opinion of the Investigator, makes the subject unsuitable for participation in the study.

Note: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 52 weeks
  Frequency of treatment-related adverse events (AEs), serious adverse events (SAEs), and changes from baseline in relevant clinical laboratory tests
Proportion of patients who can stand unassisted for at least 3 seconds at Month 12 | 52 weeks
Change from baseline on Hammersmith Functional Motor Scale - Expanded (HFMSE) scores at Month 12 | 52 weeks
  HFMSE consists of 33 activities that can be scored one of three ways: 0 for unable to perform, 1 for performs with modification/adaptation, and 2 for performs without modification.

SECONDARY OUTCOMES:
Proportion of patients treated with GC101 who achieve motor milestone of walk alone for 5 steps at Month 12 | 52 weeks

OTHER OUTCOMES:
Change from baseline in independent ventilatory support time at Month 12 | 52 weeks
Number of patients whose HFMSE scores improve more than 3 at Month 12 | 52 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking University， First Hospital, Department of Pediatrics, Beijing
  - Bayi Children's Hospital, Seventh Medical Center, PLA general hospital, Beijing
  - West China Second University Hospital, Sichuan University, Chengdu
  - Children's Hospital of Chongqing Medical University, Chongqing
  - Tongji Medical college of Huazhong University of Science&Technology, Affiliated Children's Hospital, Wuhan

IPD SHARING:
Plan to Share IPD: No